CLINICAL TRIAL: NCT02620306
Title: A Randomized, Double-blind, Active Control, Parallel Group, Titration, Multicenter Study to Evaluate the Efficacy and Safety of Fimasartan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BR-FMS-CT-303
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2021-05

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Fimasartan(A) (Experimental)
  Interventions: Drug: Fimsartan 60mg~120mg
- Fimasartan(B) (Experimental)
  Interventions: Drug: Fimsartan 60mg~120mg
- Losartan(A) (Active Comparator)
  Interventions: Drug: Losartan 50mg~100mg
- Losartan(B) (Active Comparator)
  Interventions: Drug: Losartan 50mg~100mg

INTERVENTIONS:
Drug: Fimsartan 60mg~120mg — Standard BP control group (SBP < 140 mmHg). In case of patients with blood pressure that cannot be controlled to the targeted level during the entire clinical study period, the dose of study drug is increased or other antihypertensive drugs are administered concomitantly.
  Arms: Fimasartan(A)
Drug: Fimsartan 60mg~120mg — Strict BP control group (SBP < 130 mmHg). In case of patients with blood pressure that cannot be controlled to the targeted level at each visit during the entire clinical study period, the dose of study drug is increased or other antihypertensive drugs are administered concomitantly.
  Arms: Fimasartan(B)
Drug: Losartan 50mg~100mg — Standard BP control group (SBP < 140 mmHg). In case of patients with blood pressure that cannot be controlled to the targeted level during the entire clinical study period, the dose of study drug is increased or other antihypertensive drugs are administered concomitantly.
  Arms: Losartan(A)
Drug: Losartan 50mg~100mg — Strict BP control group (SBP < 130 mmHg). In case of patients with blood pressure that cannot be controlled to the targeted level at each visit during the entire clinical study period, the dose of study drug is increased or other antihypertensive drugs are administered concomitantly.
  Arms: Losartan(B)

SUMMARY:
The purpose of this study is to evaluate the Efficacy and Safety of Fimasartan in patients with hypertensive diabetic chronic kidney disease.

DETAILED DESCRIPTION:
The randomized subjects will take the investigational product (Fimasartan or Losartan) corresponding to each treatment group for 24 weeks. After that, all subjects will take Fimasartan for additional 120 weeks in an open-label, 2-parallel group study conducted with 2 groups in accordance with the blood pressure control criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 19 years or older
2. Blood pressure: Mean blood pressure is as below at screening.

   * For treatment-naïve patients: 140 mmHg ≤ SBP < 180 mmHg and DBP < 110 mmHg
   * For patients who are taking ACEI or ARB: 130 mmHg ≤ SBP < 180 mmHg and DBP < 110 mmHg
3. eGFR: ≥ 30 ml/min/1.73 m2 within the past 6 months
4. Albuminuria (ACR) excretion volume: Meets one or more of the following conditions

   * ACR > 300 mg/g (or mg/day) within the past 12 months
   * There are at least two results of 30 ≤ ACR ≤ 300 mg/g (or mg/day) within the past 12 months and the interval between the two test is at least 12 weeks.
5. Patients with diabetes
6. Voluntarily provided a written consent to participate
7. Able to understand this study, be cooperative in the execution of the study

Exclusion Criteria:

1. Severe hypertension with mean SBP ≥ 180 mmHg or DBP ≥ 110 mmHg
2. Orthostatic hypotension with symptoms
3. Insulin dependent diabetes mellitus or uncontrolled diabetes mellitus
4. Patients on dialysis, patients with clinically significant cardiac and hepatic diseases

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
To compare and evaluate the rate of change in albuminuria | 6months

SECONDARY OUTCOMES:
The time to the first occurrence of the cardiovascular composite endpoint in accordance with the blood pressure control criteria | 36months
  Cardiovascular composite endpoint: Occurrence of myocardial infarction (MI) and stroke; hospitalization due to heart failure and unstable angina; coronary revascularization and peripheral revascularization; and all caused death
The time to the first occurrence of the renal composite endpoint in accordance with the blood pressure control criteria | 36months
  Renal composite endpoint: The time point where the reduction in eGFR of ≥ 50% compared with baseline eGFR; the time where the progression to ESRD is confirmed (in case of the initiation of long-term dialysis or renal transplantation); all caused death
The time to the first occurrence of the combined cardiovascular and renal composite endpoint in accordance with the blood pressure control criteria | 36months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park CH, Hong SJ, Kim SG, Shin SJ, Kim DK, Lee JP, Han SY, Lee S, Won JC, Kang YS, Park J, Han BG, Na KR, Hur KY, Kim YJ, Park S, Yoo TH. Blood pressure control in diabetic kidney disease: a post-hoc analysis of the FANTASTIC trial. Clin Hypertens. 2024 Aug 1;30(1):20. doi: 10.1186/s40885-024-00280-x. PMID 39085979
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Kim JY, Son JW, Park S, Yoo TH, Kim YJ, Ryu DR, Chin HJ. FimAsartaN proTeinuriA SusTaIned reduCtion in comparison with losartan in diabetic chronic kidney disease (FANTASTIC): study protocol for randomized controlled trial. Trials. 2017 Dec 29;18(1):632. doi: 10.1186/s13063-017-2375-8. PMID 29284530